CLINICAL TRIAL: NCT00232362
Title: Effect of Pioglitazone on Left Ventricular Diastolic Function in Type 2 Diabetes Mellitus
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was not conducted as the Principal Investigator left the institution
Sponsor: Texas Tech University Health Sciences Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: L05-115
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2015-04-13 (Estimated); Status verified 2015-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; Rosiglitazone

INTERVENTIONS:
Drug: Pioglitazone (Actos)
Drug: Anti-diabetic agent other than pioglitazone or rosiglitazone

SUMMARY:
This study is being done to determine if pioglitazone (Actos) is helpful to patients with type 2 diabetes and could possibly prevent harmful consequences of cardiovascular disease in diabetic patients.

DETAILED DESCRIPTION:
Cross sectional and population-based studies indicate that at least one third of all patients with congestive heart failure (CHF) have a normal or near normal ejection fraction, which is thought to be secondary to diastolic dysfunction or failure. The mortality rates among the patients with diastolic failure ranges from 5-8% annually, as compared with 10-15% among patients with systolic heart failure. The morbidity associated with diastolic heart failure is similar to that of systolic heart failure. Several studies have shown that even simple Doppler evidence of diastolic dysfunction is an independent risk factor for the development of CHF and cardiac death and increased all cause mortality. Several studies indicate that left ventricular diastolic dysfunction (LVDD) represent the earliest preclinical manifestation of diabetic cardiomyopathy that can progress to symptomatic heart failure. Recent studies have demonstrated up to 60% of asymptomatic, normotensive patients with type 2 diabetes have LVDD when assessed by conventional echocardiography including the response to the Valsalva maneuver. A recent study using conventional Doppler, valsalva maneuver, color M-mode echocardiography and tissue doppler imaging assessed the diastolic dysfunction in asymptomatic normotensive patients with diabetes mellitus and found diastolic dysfunction in about 75% of these patients. Cardiovascular disease is the leading cause of death in patients with type 2 diabetes mellitus. Although diabetic patients have a large number of cardiovascular risk factors, like hyperlipidemia and hypertension, the diabetic cardiomyopathy occurs independent of these risk factors. Recently animal models have shown that LVDD may be prevented by chronic treatment with peroxisome-proliferator-activated receptors gamma (PPAR) agonists, like thiazolidinediones, in type 2 diabetic rats. Thiazolidinediones act through PPAR, but the exact mechanism by which they improve LVDD is not known. With this background knowledge, we wanted to study the effect of Pioglitazone, which is PPAR agonist and partial PPAR agonist, on the left ventricular diastolic dysfunction in type 2 diabetic human subjects, which has not been studied so far. If this therapy proves to have beneficial effect on the LVDD it will help in preventing the deleterious consequences of diastolic dysfunction in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with type 2 diabetes mellitus (DM)
2. Ages 18 to 65 years old
3. Patients with left ventricular diastolic dysfunction (LVDD) and ejection fraction (EF) > 50%

Exclusion Criteria:

1. Patients with uncontrolled hypertension
2. Patients with active myocardial ischemia with Canadian Cardiovascular Society (CCS) > II or known coronary artery disease (CAD)
3. Patients with atrial fibrillation
4. Patients with systolic heart failure
5. Patients with mitral regurgitation grade 2 or more
6. Patients with restrictive cardiomyopathy
7. Patients with constrictive pericarditis
8. Pregnant female patients
9. Recent stroke
10. Sepsis
11. Liver enzymes more than 2.5 times the normal
12. Hemoglobin < 11g/dl or hematocrit < 30%
13. Terminal cancer
14. Patients on fibrates group of lipid lowering agents
15. Patients already on pioglitazone or rosiglitazone
16. Patients who are placed in the control group may not be currently taking a medication in the glitazones drug class.
17. Current or prior use of Pioglitazone or Rosiglitazone within the preceding 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in diastolic function parameters: early peak to late peak velocity (E/A) ratio
deceleration time (DT)
isovolumic relaxation time (IVRT)
E/A ratio percent change with Valsalva maneuver more than 40%
annular tissue Doppler velocity

CONTACTS AND LOCATIONS:
Overall Officials: Chanwit Roongsritong, MD, Principal Investigator — TTUHSC